CLINICAL TRIAL: NCT04431934
Title: Open-label, Randomized Study to Assess the Efficacy of a Probiotic or Fecal Microbiota Transplantation (FMT) on the Eradication of Rectal Multidrug-resistant Gram-negative Bacilli (MDR-GNB) Carriage (PROFTMDECOL)
Brief Title: Efficacy of a Probiotic or Fecal Microbiota Transplantation (FMT) on the Eradication of Rectal Multidrug-resistant Gram-negative Bacilli (MDR-GNB) Carriage (PROFTMDECOL)
Acronym: PROFTMDECOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, José Antonio Martinez, MD, PhD, Senior Consultor, Assistant Profesor of Medicine (University of Barcelona), Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI19/00842
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: CARRIER STATE
Keywords: fecal microbiota transplantation; probiotics; carbapenemase-producing Enterobacteriaceae; multiple-drug resistant Pseudomonas aeruginosa; ESBl-producing Klebsiella pneumoniae
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, single center, parallel-group, randomized, open-label, clinical research with non pharmacological products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention): No intervention arm
- PROBIOTIC (Active Comparator)
  Interventions: Dietary Supplement: PROBIOTIC
- FMT REGIMEN (Active Comparator)
  Interventions: Dietary Supplement: FMT REGIMEN

INTERVENTIONS:
Dietary Supplement: PROBIOTIC — Participants assigned to the probiotic arm will receive 2 sachets of "Vivomixx®" dissolved in 50 L of warm water (according to the manufacturer indications) every 12 h orally or through a nasogastric tube (in this case the tube will be flushed with 50 mL of water after the administration). The probiotic will be started 24 h after the last dose of NAA and will be administered for 14 consecutive days. Each sachet of "Vivomixx®" contains a combination of 4 Lactobacillus (L. paracasei 24733, L. acidophilus 24735, L. delbrueckii ssp bulgaricus 24734, L. plantarum 24730), 3 Bifidobacteria (B. brief 24732, B. longum 24736, B. infantis 24737), and Streptococcus thermophilus 24731 at a concentration of 450 billion (45x1010) live lyophilized bacteria per sachet.
  Arms: PROBIOTIC
Dietary Supplement: FMT REGIMEN — The FMT preparation will be administered as 2 doses, once a week, of 14-17 capsules per dose. Each dose (14-17 capsules) will contain the fecal microbiota equivalent to 50 gr of stools from a healthy donor. If the patient is carrying a nasogastric tube, the content of capsules will be decapsulized (~27 gr of powder), diluted in 50 mL of water and passed through it, followed by the administration of 50 mL of water to flush the tube. The first dose will be administered 24 h after the last dose of NAA and the second dose one week later. Whenever possible, the two doses of FMT will be originated from the same donor. According to our data done by flow cytometry and bacterial culture in three replicates, each absorbate capsule contains approximately 1.12x1010 live bacteria.
  Arms: FMT REGIMEN

SUMMARY:
The working hypothesis is that in patients who are rectal carriers of MDR-GNB (Multi drug-resistant gram negative bacilli), the rate and speed of eradication of the carrier status obtained with NAA regimens are insufficient and could be improved with additional interventions directed to restore a healthy fecal microbiota or to increase the colonization resistance by the putative beneficial activity of lactate-producing bacteria and bifidobacteria. A healthier colonic microbiota environment is expected not only to promote the eradication of the existing MDR organisms but also to hinder the subsequent recolonization and hopefully the risk of infection with gut dysbiosis -associated pathogens (MDR-GNB, C. difficile and Candida).

The principal objective of the study is To compare the decolonization efficacy at the end of the study (60 ± 7 days after randomization) of the administration of a probiotic ("Vivomixx®" 2 sachets/12h for 2 weeks) versus the administration of two doses (administered a week apart) of a fecal microbiota transplantation preparation (equivalent to 50 g of healthy donor feces) and no treatment (control arm) in patients with rectal colonization with MDRGNB (ESBL-producing Klebsiella pneumoniae, CPE and MDR/XDR (multi drug-resistant/ extensively drug-resistant Pseudomonas aeruginosa).

DETAILED DESCRIPTION:
Data Collection and Processing

Recording of data All data required for the study will be recorded in the participating center using a case report form (CRF). Completeness and plausibility checks will ensure the collection of high quality data.

A CRF for each patient will be completed by authorized personnel who must be identified and authorized in writing by the Principal Investigator before they conduct any study related tasks.

A delegation of responsibility log identifying who can enter data and/or sign off a CRF will be maintained by the Principal Investigator.

The subject's number and date of entry into the study, along with a study identifier, should be recorded in the subject's study records. The following should also be recorded in the study records: confirmation of written consent, the subject's clinical status, date of every study visit, copies of all relevant reports, comments on results and reference to serious adverse events and related adverse events.

Direct access to source data/documents Investigators will ensure access to the source documents of the staff responsible for guaranteeing data quality and data analysis. In addition, access to documentation will be provided, if necessary, to the staff duly authorized by the sponsor (study monitors).

Data management The Investigator must ensure the accuracy, completeness, legibility and timelines of data reported in the CRF and all required reports.

Archiving and storage of data The investigator is responsible for maintaining all records which enable the conduct of the study at the site to be fully documented, in accordance applicable national regulatory requirements. Timeliness and completeness of the documentation will be regularly checked by the clinical monitor. All completed study related documents (e.g. eletronic CRF, Informed consent forms, Subject identification log, etc) must be archived at site.

QUALITY CONTROL The purpose of monitoring is to verify that the rights and wellbeing of human subjects are protected; that the study is accurate, complete and verifiable with source data and that the study is conducted in compliance with the protocol, and the applicable regulatory requirements. A monitoring plan will be designed. The monitoring plan will establish the guideline for conducting all the monitoring activities. Source data will be verified during on-site monitoring visits. During the visits, the monitor will compare the data entered into the CRF with the source documents. The nature and location of all source documents will be identified to ensure that all sources of original data required to complete the eCRF are known to the monitor and study-site personnel and are accessible for verification. During monitoring visits, the relevant study-site personnel should be available, the source documentation accessible, and a suitable environment provided for review of study related documents.

Criteria for termination and /or discontinuation The participants will discontinue study participation if they are unwilling or unable to meet the protocol requirements in terms of the visit schedule or if the patient or the investigator considers it is best to end their participation in the study. All participants have the right to withdraw their consent at any time during the study without prejudice to them.

All follow-up terminations of study subjects and the reasons for them must be reported immediately to the study monitor and be duly documented both in the medical records and the case report form.

Drug accountability Drug accountability will be carried out at each study visit for those patients assigned to the Probiotic arm. FMT administration will always be performed under direct observation of one of the investigators and if ambulatory, the patient will remain under observation in the outpatient clinic during at least 2 hours after the procedure.

Source data verification Source documents are defined as all observations or notes recorded on the clinical interventions, and all reports and notes required for assessment and reconstruction of the research study.

Whenever possible the original document should be kept as the source document; however, provision of a photocopy which is clear, legible and an exact duplicate of the original document and signed by the principal investigator is acceptable.

End of the clinical research The end of the clinical research is defined as the date of the last visit of last subject undergoing the study.

Statistical analysis For the primary outcome the main analysis will be performed according to the intention to treat principle, considering as intention-to-treat population all randomized patients. Missing RS will be considered as positive. In addition, the investigators intend to do a per protocol analysis, evaluating only the patients who end the treatment and end the study. Categorical variables will be compared by the Fisher exact test and continuous ones the the student t-test or Mann-Whitney test. Univariate logistic regression with group assignment as predictor variable and clinical characteristics and decolonization as outcome will be performed to calculate OR and 95% confidence intervals. In the event of imbalance in the distribution of potential confounder despite randomization, a multivariate logistic regression analysis with decolonization as de dependent variable and group assignment as one of the explanatory variables will be carried out.

All randomised patients will be included in the "intention-to-treat population" for analysis.

Patients withdrawn for any reason or lost to follow-up will be considered as treatment failure in this analysis.

Subgroup analyses An analysis of efficacy for each bacterial species/resistance determinant (ESBL-producing K.pneumoniae, carbapenemase-producing enterobacteriaceae, MDR-P. aeruginosa) are planned

Interim analysis A safety interim analysis is planned after inclusion of the first 100 individuals in the study.

Analysis Centre Data will be analyzed in the "Institut Clinic de Medicina Interna, Dermatologia I Infeccions del Hospital Clinic de Barcelona".

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years-old).
2. Admitted to the Hospital Clinic of Barcelona with documented rectal colonization whitin the previous 7 days by rectal swabbing with MDR-GNB (ESBL-producing Klebsiella pneumoniae, carbapenemase-producing Enterobacterial (CPE) and MDR/XDR Pseudomonas aeruginosa).
3. Eligible for routine digestive decolonization (7 days oral administration of nonabsorbable antibiotics (NAA).
4. Capable to provide informed consent (by themselves or through their legal representatives).

Exclusion Criteria:

1. Pregnant women or breastfeeding.
2. Neutropenic patients (total neutrophil count <500 cell/mm3)*.
3. HIV-infected patients with CD4(cluster of differentiation 4) count <200 cell/mm3.
4. Patients with active C. difficile infection.
5. Patients with ileus or bowel obstruction.
6. Patients with documented or suspected bowel perforation.
7. Patients with a colistin-resistant MDR-GNB.

   * Solid organ or hematopoietic organ transplant recipients without neutropenia will qualify for inclusion in the study. This is based on preliminary data on the safety of probiotics without Saccharomyces boulardii/cerevisae in transplant recipients of several organs (hematopoietic precursors, liver, kidney, small intestine) and on the preliminary safety data of FMT in nonneutropenic patients with hematological disorders including hematopoietic cell transplantation (25,42,43). However, the condition of transplant recipients will be assessed inan individual basis and only those patients that by consensus with their attending physician will be judged to be at a very low risk of complications derived from the use of the probiotic o fecal microbiota will be considered for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with digestive decolonization rate | At the end of study (60 ± 7 days after the randomization).
  Proportion of patients with digestive decolonization rate defined as negative rectal swab (RS) for the target MDR-GNB (ESBL-producing Klebsiella pneumoniae, CPE and MDR/XDR Pseudomonas aeruginosa) at the end of study (60 ± 7 days after the randomization).

SECONDARY OUTCOMES:
Digestive decolonization rate defined as a negative fecal sample | At the end of study treatment (3 weeks after randomization).
  Proportion of patients with digestive decolonization rate defined as a negative fecal sample for the target MDR-GNB at the end of study treatment (3 weeks after randomization).
Digestive decolonization rate defined as a negative rectal swab | (week 1 after randomization).
  Proportion of patients with digestive decolonization rate defined as a negative rectal swab for the target MDR-GNB after the decontamination period with non-absorbable antibiotics (week 1 after randomization).
target MDR-GNB or any other MDR-GNB in any control RS or fecal sample | through study completion, an average of 1 year
  Proportion of patients with target MDR-GNB or any other MDR-GNB in any control RS or fecal sample during the study period.
clinical infections | through study completion, an average of 1 year
  Proportion of patients with clinical infections during the study period.
development of resistance to colistin or amikacin | through study completion, an average of 1 year
  Proportion of patients with development of resistance to colistin or amikacin in any strain isolated in control RS or fecal sample during the study period.
Changes in fecal microbiota composition | At the end of study treatment (3 weeks after randomization).
  Changes from baseline in fecal microbiota composition at the end of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Martinez, PhD, Principal Investigator — senior consultant; Ana del rio, PhD, Principal Investigator — senior consultant
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make individual participant data available

REFERENCES:
- [Background] Giannella M, Trecarichi EM, De Rosa FG, Del Bono V, Bassetti M, Lewis RE, Losito AR, Corcione S, Saffioti C, Bartoletti M, Maiuro G, Cardellino CS, Tedeschi S, Cauda R, Viscoli C, Viale P, Tumbarello M. Risk factors for carbapenem-resistant Klebsiella pneumoniae bloodstream infection among rectal carriers: a prospective observational multicentre study. Clin Microbiol Infect. 2014 Dec;20(12):1357-62. doi: 10.1111/1469-0691.12747. Epub 2014 Aug 11. PMID 24980276
- [Background] Amit S, Mishali H, Kotlovsky T, Schwaber MJ, Carmeli Y. Bloodstream infections among carriers of carbapenem-resistant Klebsiella pneumoniae: etiology, incidence and predictors. Clin Microbiol Infect. 2015 Jan;21(1):30-4. doi: 10.1016/j.cmi.2014.08.001. Epub 2014 Oct 12. PMID 25636924
- [Background] Girmenia C, Rossolini GM, Piciocchi A, Bertaina A, Pisapia G, Pastore D, Sica S, Severino A, Cudillo L, Ciceri F, Scime R, Lombardini L, Viscoli C, Rambaldi A; Gruppo Italiano Trapianto Midollo Osseo (GITMO); Gruppo Italiano Trapianto Midollo Osseo GITMO. Infections by carbapenem-resistant Klebsiella pneumoniae in SCT recipients: a nationwide retrospective survey from Italy. Bone Marrow Transplant. 2015 Feb;50(2):282-8. doi: 10.1038/bmt.2014.231. Epub 2014 Oct 13. PMID 25310302
- [Background] Giannella M, Bartoletti M, Morelli MC, Tedeschi S, Cristini F, Tumietto F, Pasqualini E, Danese I, Campoli C, Lauria ND, Faenza S, Ercolani G, Lewis R, Pinna AD, Viale P. Risk factors for infection with carbapenem-resistant Klebsiella pneumoniae after liver transplantation: the importance of pre- and posttransplant colonization. Am J Transplant. 2015 Jun;15(6):1708-15. doi: 10.1111/ajt.13136. Epub 2015 Mar 4. PMID 25754742
- [Background] Septimus EJ, Schweizer ML. Decolonization in Prevention of Health Care-Associated Infections. Clin Microbiol Rev. 2016 Apr;29(2):201-22. doi: 10.1128/CMR.00049-15. PMID 26817630
- [Background] Huttner B, Haustein T, Uckay I, Renzi G, Stewardson A, Schaerrer D, Agostinho A, Andremont A, Schrenzel J, Pittet D, Harbarth S. Decolonization of intestinal carriage of extended-spectrum beta-lactamase-producing Enterobacteriaceae with oral colistin and neomycin: a randomized, double-blind, placebo-controlled trial. J Antimicrob Chemother. 2013 Oct;68(10):2375-82. doi: 10.1093/jac/dkt174. Epub 2013 May 29. PMID 23719234
- [Background] Rieg S, Kupper MF, de With K, Serr A, Bohnert JA, Kern WV. Intestinal decolonization of Enterobacteriaceae producing extended-spectrum beta-lactamases (ESBL): a retrospective observational study in patients at risk for infection and a brief review of the literature. BMC Infect Dis. 2015 Oct 28;15:475. doi: 10.1186/s12879-015-1225-0. PMID 26511929
- [Background] Machuca I, Gutierrez-Gutierrez B, Perez Cortes S, Gracia-Ahufinger I, Serrano J, Madrigal MD, Barcala J, Rodriguez-Lopez F, Rodriguez-Bano J, Torre-Cisneros J. Oral decontamination with aminoglycosides is associated with lower risk of mortality and infections in high-risk patients colonized with colistin-resistant, KPC-producing Klebsiella pneumoniae. J Antimicrob Chemother. 2016 Nov;71(11):3242-3249. doi: 10.1093/jac/dkw272. Epub 2016 Jul 26. PMID 27494911
- [Background] Bar-Yoseph H, Hussein K, Braun E, Paul M. Natural history and decolonization strategies for ESBL/carbapenem-resistant Enterobacteriaceae carriage: systematic review and meta-analysis. J Antimicrob Chemother. 2016 Oct;71(10):2729-39. doi: 10.1093/jac/dkw221. Epub 2016 Jun 17. PMID 27317444
- [Background] Lubbert C, Faucheux S, Becker-Rux D, Laudi S, Durrbeck A, Busch T, Gastmeier P, Eckmanns T, Rodloff AC, Kaisers UX. Rapid emergence of secondary resistance to gentamicin and colistin following selective digestive decontamination in patients with KPC-2-producing Klebsiella pneumoniae: a single-centre experience. Int J Antimicrob Agents. 2013 Dec;42(6):565-70. doi: 10.1016/j.ijantimicag.2013.08.008. Epub 2013 Sep 19. PMID 24100228
- [Background] Tascini C, Sbrana F, Flammini S, Tagliaferri E, Arena F, Leonildi A, Ciullo I, Amadori F, Di Paolo A, Ripoli A, Lewis R, Rossolini GM, Menichetti F; GENGUT Study Group. Oral gentamicin gut decontamination for prevention of KPC-producing Klebsiella pneumoniae infections: relevance of concomitant systemic antibiotic therapy. Antimicrob Agents Chemother. 2014;58(4):1972-6. doi: 10.1128/AAC.02283-13. Epub 2014 Jan 13. PMID 24419337
- [Background] Oren I, Sprecher H, Finkelstein R, Hadad S, Neuberger A, Hussein K, Raz-Pasteur A, Lavi N, Saad E, Henig I, Horowitz N, Avivi I, Benyamini N, Fineman R, Ofran Y, Haddad N, Rowe JM, Zuckerman T. Eradication of carbapenem-resistant Enterobacteriaceae gastrointestinal colonization with nonabsorbable oral antibiotic treatment: A prospective controlled trial. Am J Infect Control. 2013 Dec;41(12):1167-72. doi: 10.1016/j.ajic.2013.04.018. PMID 24274912
- [Background] de Jonge E, Schultz MJ, Spanjaard L, Bossuyt PM, Vroom MB, Dankert J, Kesecioglu J. Effects of selective decontamination of digestive tract on mortality and acquisition of resistant bacteria in intensive care: a randomised controlled trial. Lancet. 2003 Sep 27;362(9389):1011-6. doi: 10.1016/S0140-6736(03)14409-1. PMID 14522530
- [Background] de Smet AM, Kluytmans JA, Cooper BS, Mascini EM, Benus RF, van der Werf TS, van der Hoeven JG, Pickkers P, Bogaers-Hofman D, van der Meer NJ, Bernards AT, Kuijper EJ, Joore JC, Leverstein-van Hall MA, Bindels AJ, Jansz AR, Wesselink RM, de Jongh BM, Dennesen PJ, van Asselt GJ, te Velde LF, Frenay IH, Kaasjager K, Bosch FH, van Iterson M, Thijsen SF, Kluge GH, Pauw W, de Vries JW, Kaan JA, Arends JP, Aarts LP, Sturm PD, Harinck HI, Voss A, Uijtendaal EV, Blok HE, Thieme Groen ES, Pouw ME, Kalkman CJ, Bonten MJ. Decontamination of the digestive tract and oropharynx in ICU patients. N Engl J Med. 2009 Jan 1;360(1):20-31. doi: 10.1056/NEJMoa0800394. PMID 19118302
- [Background] Oostdijk EA, Smits L, de Smet AM, Leverstein-van Hall MA, Kesecioglu J, Bonten MJ. Colistin resistance in gram-negative bacteria during prophylactic topical colistin use in intensive care units. Intensive Care Med. 2013 Apr;39(4):653-60. doi: 10.1007/s00134-012-2761-3. Epub 2012 Dec 1. PMID 23203301
- [Background] Oostdijk EAN, Kesecioglu J, Schultz MJ, Visser CE, de Jonge E, van Essen EHR, Bernards AT, Purmer I, Brimicombe R, Bergmans D, van Tiel F, Bosch FH, Mascini E, van Griethuysen A, Bindels A, Jansz A, van Steveninck FAL, van der Zwet WC, Fijen JW, Thijsen S, de Jong R, Oudbier J, Raben A, van der Vorm E, Koeman M, Rothbarth P, Rijkeboer A, Gruteke P, Hart-Sweet H, Peerbooms P, Winsser LJ, van Elsacker-Niele AW, Demmendaal K, Brandenburg A, de Smet AMGA, Bonten MJM. Effects of decontamination of the oropharynx and intestinal tract on antibiotic resistance in ICUs: a randomized clinical trial. JAMA. 2014 Oct 8;312(14):1429-1437. doi: 10.1001/jama.2014.7247. PMID 25271544
- [Background] Wittekamp BH, Plantinga NL, Cooper BS, Lopez-Contreras J, Coll P, Mancebo J, Wise MP, Morgan MPG, Depuydt P, Boelens J, Dugernier T, Verbelen V, Jorens PG, Verbrugghe W, Malhotra-Kumar S, Damas P, Meex C, Leleu K, van den Abeele AM, Gomes Pimenta de Matos AF, Fernandez Mendez S, Vergara Gomez A, Tomic V, Sifrer F, Villarreal Tello E, Ruiz Ramos J, Aragao I, Santos C, Sperning RHM, Coppadoro P, Nardi G, Brun-Buisson C, Bonten MJM. Decontamination Strategies and Bloodstream Infections With Antibiotic-Resistant Microorganisms in Ventilated Patients: A Randomized Clinical Trial. JAMA. 2018 Nov 27;320(20):2087-2098. doi: 10.1001/jama.2018.13765. PMID 30347072
- [Background] Shayto RH, Abou Mrad R, Sharara AI. Use of rifaximin in gastrointestinal and liver diseases. World J Gastroenterol. 2016 Aug 7;22(29):6638-51. doi: 10.3748/wjg.v22.i29.6638. PMID 27547007
- [Background] Maziade PJ, Pereira P, Goldstein EJ. A Decade of Experience in Primary Prevention of Clostridium difficile Infection at a Community Hospital Using the Probiotic Combination Lactobacillus acidophilus CL1285, Lactobacillus casei LBC80R, and Lactobacillus rhamnosus CLR2 (Bio-K+). Clin Infect Dis. 2015 May 15;60 Suppl 2:S144-7. doi: 10.1093/cid/civ178. PMID 25922400
- [Background] Crum-Cianflone NF, Sullivan E, Ballon-Landa G. Fecal microbiota transplantation and successful resolution of multidrug-resistant-organism colonization. J Clin Microbiol. 2015 Jun;53(6):1986-9. doi: 10.1128/JCM.00820-15. Epub 2015 Apr 15. PMID 25878340
- [Background] Manges AR, Steiner TS, Wright AJ. Fecal microbiota transplantation for the intestinal decolonization of extensively antimicrobial-resistant opportunistic pathogens: a review. Infect Dis (Lond). 2016 Aug;48(8):587-92. doi: 10.1080/23744235.2016.1177199. Epub 2016 May 19. PMID 27194400
- [Background] Davido B, Salomon J, Lawrence C, Duran C, Batista R, de Truchis P, Dinh A. Impact of Fecal Microbiota Transplantation for Decolonization of Multidrug-Resistant Organisms May Vary According to Donor Microbiota. Clin Infect Dis. 2018 Apr 3;66(8):1316-1317. doi: 10.1093/cid/cix963. No abstract available. PMID 29272347
- [Background] Saha S, Tariq R, Tosh PK, Pardi DS, Khanna S. Faecal microbiota transplantation for eradicating carriage of multidrug-resistant organisms: a systematic review. Clin Microbiol Infect. 2019 Aug;25(8):958-963. doi: 10.1016/j.cmi.2019.04.006. Epub 2019 Apr 12. PMID 30986562
- [Background] Bilinski J, Grzesiowski P, Sorensen N, Madry K, Muszynski J, Robak K, Wroblewska M, Dzieciatkowski T, Dulny G, Dwilewicz-Trojaczek J, Wiktor-Jedrzejczak W, Basak GW. Fecal Microbiota Transplantation in Patients With Blood Disorders Inhibits Gut Colonization With Antibiotic-Resistant Bacteria: Results of a Prospective, Single-Center Study. Clin Infect Dis. 2017 Aug 1;65(3):364-370. doi: 10.1093/cid/cix252. PMID 28369341
- [Background] Huttner BD, de Lastours V, Wassenberg M, Maharshak N, Mauris A, Galperine T, Zanichelli V, Kapel N, Bellanger A, Olearo F, Duval X, Armand-Lefevre L, Carmeli Y, Bonten M, Fantin B, Harbarth S; R-Gnosis WP3 study group. A 5-day course of oral antibiotics followed by faecal transplantation to eradicate carriage of multidrug-resistant Enterobacteriaceae: a randomized clinical trial. Clin Microbiol Infect. 2019 Jul;25(7):830-838. doi: 10.1016/j.cmi.2018.12.009. Epub 2019 Jan 4. PMID 30616014
- [Background] Tariq R, Pardi DS, Bartlett MG, Khanna S. Low Cure Rates in Controlled Trials of Fecal Microbiota Transplantation for Recurrent Clostridium difficile Infection: A Systematic Review and Meta-analysis. Clin Infect Dis. 2019 Apr 8;68(8):1351-1358. doi: 10.1093/cid/ciy721. PMID 30957161

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04431934/Prot_SAP_000.pdf